CLINICAL TRIAL: NCT01155362
Title: A Phase 2a, Randomized, Double Blind, Placebo Controlled, Multi-Center Study to Evaluate the Safety and Efficacy of Intravenous Infusion of Human Placenta-Derived Cells (PDA001) for the Treatment of Adults With Moderate-to-Severe Crohn's Disease
Brief Title: A Multi-Center Study to Evaluate the Safety and Efficacy of Intravenous Infusion of Human Placenta-Derived Cells (PDA001) for the Treatment of Adults With Moderate-to-Severe Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celularity Incorporated (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCT-PDA001-002
Record Dates: First submitted 2010-05-26; First posted 2010-07-01 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2014-07

CONDITIONS: Crohn's Disease
Keywords: Human Placenta-Derived Cells for the Treatment of Moderate-to-Severe Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 unit Human Placenta-Derived Cells PDA001 (Experimental): 1 unit PDA001 in 240 millilters (mL) infused intravenously in one arm on Day 0 and Day 7.
  Interventions: Biological: Human Placenta-Derived Cells PDA001 Intravenous Infusion
- 4 units Human Placenta-Derived Cells PDA001 (Experimental): 4 units PDA001 in 240 mL infused intravenously in one arm on Day 0 and Day 7.
  Interventions: Biological: Human Placenta-Derived Cells PDA001 Intravenous Infusion
- vehicle control (Placebo Comparator): 4 units placebo in 240 mL infused intravenously in one arm on Day 0 and Day 7.
  Interventions: Drug: Vehice Control
- 8 units Human Placenta-Derived Cells PDA001 (Experimental): 4 units PDA-001 in 240 mL infused intravenously in each arm on Day 0 and Day 7 or 8 units PDA-001 in 240 mL infused intravenously in one arm on Day 0 and Day 7
  Interventions: Biological: Human Placenta-Derived Cells PDA001 Intravenous Infusion

INTERVENTIONS:
Biological: Human Placenta-Derived Cells PDA001 Intravenous Infusion
  Arms: 1 unit Human Placenta-Derived Cells PDA001; 4 units Human Placenta-Derived Cells PDA001; 8 units Human Placenta-Derived Cells PDA001
Drug: Vehice Control
  Other Names: Placebo
  Arms: vehicle control

SUMMARY:
The primary objective of the study is to estimate the treatment effect of PDA001 (evaluating 3 different PDA001 dosings) versus placebo in subjects with moderate-to-severe Crohn's Disease. The secondary objective of the study is to assess the safety and tolerability of PDA001 versus placebo in the above-mentioned patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 18-75 years
2. Understand and voluntarily sign an informed consent
3. Able to adhere to the study visit schedule and other protocol requirements
4. Minimum weight of 50 kg
5. A female of childbearing potential (FCBP)† must have a negative urine pregnancy test at screening (Visit 1) and immediately prior to all doses of IP. In addition, sexually active FCBP must agree to use two of the adequate forms of contraception methods for the duration of the study and the follow-up period. A FCBP must agree to have pregnancy tests at least every 4 weeks during the study. Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in reproductive sexual activity with FCBP for the duration of the study and the follow-up period.
6. Subject must have inflammatory CD 6 months prior to treatment and have confirmation of ongoing disease activity by colonoscopy or (other method) at screening
7. Subject must have a CDAI score > 220 and < 450 as assessed between Visit 1 and Visit 2
8. The Subject must have failed, i.e., had an inadequate response or lost response (recurrence of symptoms) to an agent, or documented intolerance to an agent at any time

Exclusion Criteria:

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
2. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study

A female of childbearing potential is a sexually mature woman who:

1. has not undergone a hysterectomy or bilateral oophorectomy
2. has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2012-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
A reduction from baseline by 25% and/or > 100 points in the Crohn's Disease Activity Index (CDAI) scores at both Week 4 (Day 29) and at Week 6 (Day 43). | Week 4 (Day 29) and Week 6 (Day 43)
  Crohn's disease activity index (CDAI) responders are subjects achieving either clinical response (a reduction in CDAI score of ≥100 points from Week 0), or remission (CDAI ≤150). CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease.

SECONDARY OUTCOMES:
The induction of a clinical remission defined as a Crohn's Disease Activity Index score of < 150 points at both Week 4 (Day 29) and Week 6 (Day 43) | Week 4 (Day 29) and Week 6 (Day 43)
  Crohn's disease activity index (CDAI) is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: Solveig Ericson, MD, Study Director — Celularity Incorporated
Locations (13):
- United States (13):
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California, Irvine, Orange, California
  - Yale School of Medicine Digestive Diseases, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Mt Sinai Hospital, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Stony Brook University, Stony Brook, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - McGuire VA Medical Center, Richmond, Virginia